CLINICAL TRIAL: NCT06348602
Title: Evaluation of Safety and Efficacy for the Prevention of Ocular Graft-versus-host Disease With Ophthalmic Tacrolimus vs. Ophthalmic Cyclosporine in Non-myeloablative Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: Evaluation of Safety & Efficacy for the Prevention of Ocular GVHD With Ophthalmic Tacrolimus vs Cyclosporine in Allo-HSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Hematology, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI23-00201
Record Dates: First submitted 2023-10-30; First posted 2024-04-04 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Ocular Graft-versus-host Disease
Keywords: Allogeneic; Hematopoietic Stem Cell Transplantation; Dry eye syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Experimental, prospective, randomized, unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical cyclosporine (Active Comparator): Topical cyclosporine ophthalmic solution 0.1%, with a dosage of 1 drop in each eye every 12 hours, continued for a duration of 12 continuous months.
  Composition: Each ml contains Cyclosporine A 0.1% w/v (1 mg/ml) in a sterile aqueous vehicle q.s.
  Interventions: Drug: Cyclosporine ophthalmic solution 0.1%
- Topical tacrolimus (Experimental): Topical tacrolimus ophthalmic ointment 0.03%, with a dosage of approximately 1 cm or the necessary amount to cover the lower fornix, every 12 hours, continued for a duration of 12 continuous months Composition: Each gram contains Tacrolimus 0.03% w/w (0.3 mg/g) in a sterile ointment base q.s.
  Interventions: Drug: Tacrolimus ophthalmic ointment 0.03%

INTERVENTIONS:
Drug: Cyclosporine ophthalmic solution 0.1% — Ophthalmic prophylaxis begins once engraftment is documented, with a dose of 1 drop in each eye every 12 hours, continued for a duration of 12 continuous months
  Arms: Topical cyclosporine
Drug: Tacrolimus ophthalmic ointment 0.03% — Ophthalmic prophylaxis begins once engraftment is documented, with a dose of approximately 1 cm or the necessary amount to cover the lower fornix, every 12 hours, continued for a duration of 12 continuous months
  Arms: Topical tacrolimus

SUMMARY:
Chronic GVHD (cGVHD) is a predominant cause of mortality and disability not related to relapse; it occurs in 30 to 70% of patients. The majority of patients with cGVHD present with ocular involvement with a reported incidence of 40-60%. Symptoms can range from mild dry eye syndrome to severe epithelial defects that can generate corneal perforation and loss of vision. The most accepted pharmacological modality is the topical application of cyclosporine A; on the other hand, tacrolimus has shown greater immunosuppressive power when used in ocular GVHD. However, this effectiveness is limited since by the time the manifestations appear, there is already permanent damage to the lacrimal gland due to the lymphocytic infiltration; so it is necessary to use a prevention strategy before these manifestations appear. Previously, the employment of ocular cyclosporine drops as ocular GVHD prophylaxis was assessed to evaluate safety and effectiveness, showing that it is well tolerated and can limit the appearance of severe dry eye manifestations in a small group of patients. The purpose of this work is to compare the two modalities currently accepted for the treatment of the disease, but in a prophylactic way; topical ciclosporin A against topical tacrolimus, to determine the safety and efficiency of each of them as a preventive measure to limit the risk of developing the appearance of ocular cGVHD and the permanent consequences that this generates.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be assigned a participant number to anonymize their data and collect information, including age, sex, diagnosis, stage of disease, type of procedure, and conditioning chemotherapy. Additionally, an ophthalmology evaluation will be conducted in the Ophthalmology Department of the University Hospital of the U.A.N.L. by the study team of ophthalmologists, following a standardized method and using a worksheet for dry eye and ocular surface evaluation.

Participants will be randomized to receive either treatment arm A (cyclosporine eye drops) or treatment arm B (tacrolimus ointment) through a stratified method. After the hematopoietic stem cell transplant (HSCT), information will be collected, such as the transplant details (e.g., number of cluster of differentiation 34 [CD34] cells infused, cell source, and any complications during the procedure) and medications used for the systemic GVHD prophylaxis, as well as the graft date. In addition to the standard systemic management protocol for GVHD prevention of the transplant program of the Hematology Service of the Hospital University U.A.N.L. cyclosporine or tacrolimus will be administered to participants once grafting is demonstrated, defined as the presence in the blood count of a neutrophil count that is equal to or greater than to 500/mm3 and platelet count equal to or greater than 20,000/mm3.

* Treatment arm A: topical cyclosporine 0.1% ocular drops, twice daily, one drop in each eye, with a 12-hour difference between each dose, for 12 continuous months. The commercial presentation that we will use has the following formula: Each milliliter of 0.1% solution contains Cyclosporine A 10 mg, c.b.p 1.0 ml.
* Treatment arm B: tacrolimus ointment, to be applied approximately 1cm or the amount to cover the lower fornix twice a day in each eye, with a difference of 12 hours between each dose, for 12 continuous months. The presentation of the medicine in ointment has a 10 gr tube with 0.03% drug.

Ophthalmological evaluations will be carried out at the initial visit (before the bone marrow transplant) and scheduled subsequent visits: at the time of transplant graft (variable depending on the type of transplant, between days +10 and +21 approximately), and 3, 6, 9, and 12 months from the start of treatment (day of graft). Also, they will be evaluated during all follow-up visits to the transplant department of the Hematology Service, assessing adherence and tolerance to the medication through direct questioning. The severity of ocular GVHD will be established based on the NIH criteria and the severity criteria of the international consensus on the severity of chronic ocular GVHD (ICCGVHD)

Ophthalmological variables to be evaluated

* Tear breakup time, Schirmer's test, esthesiometry, Keratograph 5M Topographer Dry Eye Assessment, upper and lower tarsus Meibomian Gland imaging (Keratograph 5M), tear osmolarity, metalloproteinase 9 levels in tears.
* Corneal and conjunctival staining measured with the Oxford Scale and the Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Scale and SICCA Ocular Staining Score (OSS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing allogeneic HSCT.
2. Patients 18 years of age or older.
3. Patients who agree to participate in the study and sign the informed consent document.

Exclusion Criteria:

1. Patients undergoing HSCT who do not continue their evaluation and follow-up in the Hematology Service of the University Hospital.
2. Patients under 18 years of age.
3. Patients who do not agree to participate in the study.
4. Patients diagnosed with previous rheumatic disease.
5. Patients with dermatological conditions undergoing systemic treatment.
6. Patients with uncontrolled thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular graft-versus-host disease in patients undergoing allo-HSCT receiving topical prophylaxis with Cyclosporine A or Tacrolimus as assessed by the International Consensus Criteria on chronic ocular graft-versus-host disease. | 2.5 years
  Severity based on an aggregate of scores of the following parameters: Schirmer's test [mm] (0, >15; 1, 11-15; 2, 6-10; 3, ≤5), Corneal fluorescein staining [points] (0, 0; 1, <2; 2, 2-3; 3, ≥4), Ocular Surface Disease Index [points] (0, <13; 1, 13-22; 2, 23-32; 3, ≥33), Conjunctival injection [points] (0, None; 1, Mild/Moderate; 2, Severe). Graded as none (0-4 points), mild/moderate (5-8 points) and severe (9-11 points), where higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Incidence of ocular graft-versus-host disease in patients undergoing allo-HSCT receiving topical prophylaxis with Cyclosporine A or Tacrolimus as assessed by the National Institutes of Health Consensus Development Projects on Chronic GVHD scoring system. | 2.5 years
  Severity graded from 0 to 3 as follows: 0: No symptoms; 1: mild dry eye symptoms not affecting activity of daily living (requiring eye drops ≤3 x per day); 2: Moderate dry eye symptoms partially affecting activity of daily living (requiring eye drops >3 x per day or punctal plugs) WITHOUT new vision impairment due to keratoconjunctivitis sicca; 3: Severe dry eye symptoms significantly affecting activity of daily living (special eyewear to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to keratoconjunctivitis sicca. Note: higher scores mean a worse outcome.
Prevalence of ocular GVHD based on historical records in the hematology service of the University Hospital U.A.N.L. in patients without prophylactic treatment as assessed by the International Consensus Criteria on chronic ocular graft-versus-host disease | 10 years
  Severity based on an aggregate of scores of the following parameters: Schirmer's test [mm] (0, >15; 1, 11-15; 2, 6-10; 3, ≤5), Corneal fluorescein staining [points] (0, 0; 1, <2; 2, 2-3; 3, ≥4), Ocular Surface Disease Index [points] (0, <13; 1, 13-22; 2, 23-32; 3, ≥33), Conjunctival injection [points] (0, None; 1, Mild/Moderate; 2, Severe). Graded as none (0-4 points), mild/moderate (5-8 points) and severe (9-11 points), where higher scores mean a worse outcome.
Severity of ocular GVHD based on historical records in the hematology service of the University Hospital U.A.N.L. in patients without prophylactic treatment, as assessed by the International Consensus Criteria on chronic ocular graft-versus-host disease. | 10 years
  Severity based on an aggregate of scores of the following parameters: Schirmer's test [mm] (0, >15; 1, 11-15; 2, 6-10; 3, ≤5), Corneal fluorescein staining [points] (0, 0; 1, <2; 2, 2-3; 3, ≥4), Ocular Surface Disease Index [points] (0, <13; 1, 13-22; 2, 23-32; 3, ≥33), Conjunctival injection [points] (0, None; 1, Mild/Moderate; 2, Severe). Graded as none (0-4 points), mild/moderate (5-8 points) and severe (9-11 points), where higher scores mean a worse outcome.
Prevalence of ocular GVHD based on historical records in the hematology service of the University Hospital U.A.N.L. in patients without prophylactic treatment, as assessed by the National Institutes of Health Consensus on Chronic GVHD scoring system. | 10 years
  Severity graded from 0 to 3 as follows: 0: No symptoms; 1: mild dry eye symptoms not affecting activity of daily living (requiring eye drops ≤3 x per day); 2: Moderate dry eye symptoms partially affecting activity of daily living (requiring eye drops >3 x per day or punctal plugs) WITHOUT new vision impairment due to keratoconjunctivitis sicca; 3: Severe dry eye symptoms significantly affecting activity of daily living (special eyewear to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to keratoconjunctivitis sicca. Note: higher scores mean a worse outcome.
Severity of ocular GVHD based on historical records in the hematology service of the University Hospital U.A.N.L. in patients without prophylactic treatment, as assessed by the National Institutes of Health Consensus on Chronic GVHD scoring system. | 10 years
  Severity graded from 0 to 3 as follows: 0: No symptoms; 1: mild dry eye symptoms not affecting activity of daily living (requiring eye drops ≤3 x per day); 2: Moderate dry eye symptoms partially affecting activity of daily living (requiring eye drops >3 x per day or punctal plugs) WITHOUT new vision impairment due to keratoconjunctivitis sicca; 3: Severe dry eye symptoms significantly affecting activity of daily living (special eyewear to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to keratoconjunctivitis sicca. Note: higher scores mean a worse outcome.
Number of participants requiring adjuvant treatment for ocular GVHD in patients receiving prophylactic tacrolimus or cyclosporine for ocular GVHD. | 2.5 years
  e.g topical corticosteroids
Prevalence of Dry Eye Disease prior to the HSCT. | 2.5
  Evaluation of dry eye symptoms with the ocular surface disease index (OSDI), National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25), tear breakup time, schirmer test.
Subtypes of Dry Eye Disease prior to the HSCT | 2.5
  Evaluation of dry eye symptoms with the ocular surface disease index (OSDI), National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25), tear breakup time, schirmer test.
Number of participants requiring adjuvant treatments for the Dry Eye Disease | 2.5 years
  e.g.eye lubricant, artificial tears, autologous serum or autologous platelet-rich plasma in drops.
Incidence of other manifestations of acute and chronic GVHD, local or systemic, in patients receiving prophylactic treatment for ocular GVHD. | 2.5 years
  With The National Institutes of Health (NIH) consensus criteria used to diagnose GVHD
Number of participants with topical tacrolimus related adverse events as assessed by a questionnaire for evaluation of adverse drug events | 1 year
  Variables: frequency and severity (0-100) of burning sensation, pain, itching, discomfort, blurred vision, foreign body sensation, others.
Number of participants with topical cyclosporine related adverse events as assessed by a questionnaire for evaluation of adverse drug events | 1 year
  Variables: frequency and severity (0-100) of burning sensation, pain, itching, discomfort, blurred vision, foreign body sensation, others.

OTHER OUTCOMES:
Incidence of ocular GVHD in patients receiving prophylactic treatment for ocular GVHD. | 2.5 years
  Assessed by the Ocular Graft Versus Host Disease diagnostic criteria and grading scale according to the NIH criteria 2014 and the International Consensus Criteria on chronic ocular graft versus host disease (ICCGVHD)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de la U.A.N.L., Nuevo León, Monterrey, Mexico

REFERENCES:
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Result] Cantu-Rodriguez OG, Vazquez-Mellado A, Gonzalez-Trevino JL, Martinez-Garza DM, Gomez-De Leon A, Hawing-Zarate JA, Jaime-Perez JC, Gutierrez-Aguirre CH, Garza-Acosta AC, Mancias-Guerra C, Gonzalez-Llano O, Gonzalez-Cantu GA, Herrera-Rojas MA, Sada-Ovalle I, Gomez-Almaguer D. Cyclosporine A for the Prevention of Ocular Graft versus Host Disease in Allogeneic Hematopoietic Stem Cell Transplant Recipients Is Safe and Feasible. Acta Haematol. 2020;143(5):425-431. doi: 10.1159/000502405. Epub 2019 Sep 10. PMID 31505491
- [Result] Jung JW, Lee YJ, Yoon SC, Kim TI, Kim EK, Seo KY. Long-term result of maintenance treatment with tacrolimus ointment in chronic ocular graft-versus-host disease. Am J Ophthalmol. 2015 Mar;159(3):519-27.e1. doi: 10.1016/j.ajo.2014.11.035. Epub 2014 Dec 9. PMID 25498356
- See also: Multicenter prospective validation study for international chronic ocular graft-versus-host disease consensus diagnostic criteria — https://keio.elsevierpure.com/en/publications/multicenter-prospective-validation-study-for-international-chroni